CLINICAL TRIAL: NCT04677205
Title: Molecular Signature From Tumor to Lymph Nodes: How to Identify the Right Candidate for IIIA-N2 Lung Cancer Surgery?
Brief Title: Molecular Signature From Tumor to Lymph Nodes
Acronym: N2-3S
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Cancer Institute, France (Other Government); Ministry of Health, France (Other Government); Université de Paris (Unknown)
Responsible Party: Sponsor
Other Study IDs: D20180155; D20180155 (Other: Assistance Publique - Hôpitaux de Paris); 2019-A02635-52 (Other: N° IDRCB)
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Lung Cancer; Stage IIIA-cN2; Operated With Curative Intent; Primary Tumor Tissue Available; Node Tumor Tissue Available
Keywords: NSCLC; N2; molecular profile; prognosis
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Tumor DNA, Tumor RNA, cell free DNA from blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mediastinal lymph node (LN) involvement (N2) in non-small cell lung cancer (NSCLC) concerns 15% of resectable tumors and is associated with a poor prognosis and an overall survival reaching 9 to 49%. Literature fails to provide any definitive consensus regarding the management of these patients, except for the platinum-based doublet chemotherapy. The N2 involvement remains a matter of debate because of its not yet well-classified heterogeneity. Regarding anatomy, the Mountain and Dresler's regional LN classification for lung cancer staging remains the reference. Different studies classified IIIA-N2 disease into 4 groups, in addition to the skip-N2 phenomenon: minimal-N2, N2 single station, N2 multiple stations, and bulky-N2. Other subgroups were recently proposed for the 8th edition of the TNM: N2a1 - single station skip, N2a2 - single station non-skip, N2b - multiple stations.

The French National Cancer Institute (INCa) proposed guidelines, but in case of cN2 staging without mediastinal infiltration, guidelines remained imprecise ("resectability should be discussed for each case") and suggested surgery first, or induction chemotherapy, or concomitant chemoradiation.

Thus, optimal management of cIIIA-N2 remains controversial but complete tumor resection can be related to long-term survival in some patients, including 10 years after surgery [1]. In this situation, the identification of markers that will help select IIIA-N2 patients who will benefit from surgical resection is mandatory.

DETAILED DESCRIPTION:
We planned a comprehensive molecular characterization of tumors and lymph nodes to evaluate the impact of molecular signatures and molecular heterogeneity on disease-free survival after surgery in IIIA-N2 NSCLC patients. Identification of specific molecular profiles in primary tumors and evolution profiles in nodes might provide clues to the potential risk of metastatic evolution and trigger specific management.

For patients included prospectively, we planned to analyze cell free circulating tumor DNA (ctDNA) as prognostic marker. Because multiple biopsies are not always available in care settings, ctDNA could also be analyzed as a surrogate marker of molecular heterogeneity. Next generation sequencing (NGS) that was validated in our lab to screen ctDNA using a specific bio-informatics workflow allows accurate and cost effective ctDNA screening

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, men and women age >18 years
* Patients operated with a curative intent for an IIIA-cN2 NSCLC
* Social security affiliation
* Written informed consent for patient included in part 2 (prospective) or not opposing the use of this data for patient included in part 1 (retrospective)

Exclusion Criteria:

* Patient with T4, R1 or R2 surgical resection, sublobar resection, no radical lymphadenectomy
* Patient under protectives measures
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 230 patients in 11 French centers in order to have 200 eligible patients. Objectives are 120 patients recruited retrospectively and 110 prospectively.
  Inclusion criteria are: all consecutive patients operated with a curative intent for an IIIA-cN2 NSCLC.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival | 3 years
  To identify a molecular signature based on a comprehensive molecular analysis at genomic and transcriptomic levels linked to 3-year disease-free survival in resected IIIA-N2 NSCLC.

SECONDARY OUTCOMES:
5-year disease-free survival | 5 years
  To identify a molecular signature based on a comprehensive molecular analysis at genomic and transcriptomic levels linked to 5-year disease-free survival in resected IIIA-N2 NSCLC.
pathological architectural patterns WHO 2015 classification | 5 years
  To evaluate the impact of the pathological architectural patterns WHO 2015 classification on the 5-year cancer-specific survival and the 5-year overall survival
anatomical lymphatic spread | at the end of molecular analyses
  To identify tumor molecular patterns associated with specific anatomical lymphatic spread subgroups.
ctDNA | 3 years
  To assess ctDNA prognostic impact, before and after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Helene BLONS, PharmD PhD, Principal Investigator — Hôpital Européen Georges-Pompidou
Locations (12):
- France (12):
  - Hôpital du Haut-Lévêque, CHU de Bordeaux, Bordeaux
  - Hôpital Militaire Percy, Clamart
  - Hôpital Nord, Marseille
  - Hôpital Pasteur, CHU de Nice, Nice
  - Hegp-Aphp, Paris
  - Hôpital Européen Georges-Pompidou, Paris
  - Hôpital Bichat, Paris
  - Hôpital Cochin, Paris
  - Hôpital Pontchaillou, CHU de Rennes, Rennes
  - Hôpitaux universitaires de Strasbourg, Strasbourg
  - Hôpital Larrey, CHU de Toulouse, Toulouse
  - CHRU de Tours, Tours

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization. Processing of shared data must comply with European General Data Protection Regulation (GDPR).

REFERENCES:
- [Background] Altman DG, McShane LM, Sauerbrei W, Taube SE. Reporting recommendations for tumor marker prognostic studies (REMARK): explanation and elaboration. BMC Med. 2012 May 29;10:51. doi: 10.1186/1741-7015-10-51. PMID 22642691
- [Background] Legras A, Mordant P, Arame A, Foucault C, Dujon A, Le Pimpec Barthes F, Riquet M. Long-term survival of patients with pN2 lung cancer according to the pattern of lymphatic spread. Ann Thorac Surg. 2014 Apr;97(4):1156-62. doi: 10.1016/j.athoracsur.2013.12.047. Epub 2014 Feb 26. PMID 24582052
- [Background] Lin IF, Chang WP, Liao YN. Shrinkage methods enhanced the accuracy of parameter estimation using Cox models with small number of events. J Clin Epidemiol. 2013 Jul;66(7):743-51. doi: 10.1016/j.jclinepi.2013.02.002. Epub 2013 Apr 6. PMID 23566374
- [Background] Pecuchet N, Rozenholc Y, Zonta E, Pietrasz D, Didelot A, Combe P, Gibault L, Bachet JB, Taly V, Fabre E, Blons H, Laurent-Puig P. Analysis of Base-Position Error Rate of Next-Generation Sequencing to Detect Tumor Mutations in Circulating DNA. Clin Chem. 2016 Nov;62(11):1492-1503. doi: 10.1373/clinchem.2016.258236. Epub 2016 Sep 13. PMID 27624137
- [Background] Peduzzi P, Concato J, Feinstein AR, Holford TR. Importance of events per independent variable in proportional hazards regression analysis. II. Accuracy and precision of regression estimates. J Clin Epidemiol. 1995 Dec;48(12):1503-10. doi: 10.1016/0895-4356(95)00048-8. PMID 8543964
- [Background] Tapak L, Saidijam M, Sadeghifar M, Poorolajal J, Mahjub H. Competing risks data analysis with high-dimensional covariates: an application in bladder cancer. Genomics Proteomics Bioinformatics. 2015 Jun;13(3):169-76. doi: 10.1016/j.gpb.2015.04.001. Epub 2015 Apr 20. PMID 25907251
- [Background] Um SW, Joung JG, Lee H, Kim H, Kim KT, Park J, Hayes DN, Park WY. Molecular Evolution Patterns in Metastatic Lymph Nodes Reflect the Differential Treatment Response of Advanced Primary Lung Cancer. Cancer Res. 2016 Nov 15;76(22):6568-6576. doi: 10.1158/0008-5472.CAN-16-0873. Epub 2016 Sep 13. PMID 27634761
- [Background] Vittinghoff E, McCulloch CE. Relaxing the rule of ten events per variable in logistic and Cox regression. Am J Epidemiol. 2007 Mar 15;165(6):710-8. doi: 10.1093/aje/kwk052. Epub 2006 Dec 20. PMID 17182981